CLINICAL TRIAL: NCT04720924
Title: Computer-aided Real-time Automatic Quality-control System for Detection of Early Cancer and Precancerous Lesions on Upper Gastrointestinal Tract: a Multicenter Randomized Controlled Study
Brief Title: AQCS for Detection of Early Cancer and Precancerous Lesions on Upper Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Binzhou Medical University (Other); Shengli Oilfield Hospital (Other); Peking University Care Luzhong Hospital (Other); Linyi People's Hospital (Other); Zibo Municipal Hospital (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020SDU-QILU-1022
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Esophagogastroduodenoscopy
Keywords: Esophagogastroduodenoscopy; Gastric Cancer; esophageal cancer; Artificial Intelligence; Quality-control
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AQCS-aided group (Experimental): Patients in AQCS-aided group will go through white light EGD examination with assistance of AQCS.
  Interventions: Device: Computer-aided Real-time Automatic Quality-control System
- Control group (No Intervention): Patients in control group will go through white light EGD examination without AQCS.

INTERVENTIONS:
Device: Computer-aided Real-time Automatic Quality-control System — EGD automatic quality-control system(AQCS),developed based on deep convolutional neural network (DCNN) models,could facilitate real-time detection of upper gastrointestinal lesions, assess inspection completeness and mucosal visibility, and calculate time of EGD procedure.
  Arms: AQCS-aided group

SUMMARY:
The purpose of our study was to assess the performance of esophagogastroduodenoscopy automatic quality-control system in real-time quality control of EGD.

DETAILED DESCRIPTION:
Investigators developed a real-time quality control system of esophagogastroduodenoscopy(EGD) named EGD automatic quality-control system (AQCS). Investigators carried a prospective multicenter randomized controlled trial to assess the performance of this system in quality control of real-time EGD, including detecting the early upper gastrointestinal cancer and precancerous lesions, assessing inspection completeness, mucosal visibility, time of EGD procedure and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 years old
* Patients scheduled for white light EGD examination with anaesthesia
* American Society of Anesthesiology risk class 1, 2 or 3

Exclusion Criteria:

* Patients with known advanced esophageal or gastric cancer
* Patients with a history of esophageal or gastric surgery
* Patients scheduled for therapeutic EGD
* Patients with stenosis or obstruction of upper gastrointestinal tract
* Patients with a history of serious anesthesia-related complications
* Patients in pregnancy or lactation phase
* Patients refused to sign the informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1840 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of early cancer and precancerous lesions on upper gastrointestinal tract confirmed by pathological examination | 6 months
  The primary outcome is the detection rate of early cancer and precancerous lesions on upper gastrointestinal tract confirmed by pathological examination per group.

SECONDARY OUTCOMES:
Detection rate of early cancer and precancerous lesions on upper gastrointestinal tract in tertiary hospitals and secondary hospitals. | 6 months
  Effect of detection rate of early cancer and precancerous lesions on upper gastrointestinal tract from tertiary hospitals and secondary hospitals with assistance of AQCS.
Mean inspection completeness of two groups. | 6 months
  Inspection completeness includes taking standard images of each parts of esophageal and gastric cavity.
Mean inspection time of EGD procedure of two groups. | During procedure
  Inspection time of EGD procedure is the time endoscopy inserting to withdrawing the mouth and does not include the time of biopsy.
Detection rate of early cancer and precancerous lesions on upper gastrointestinal tract from senior, intermediate and primary endoscopist with assistance of AQCS. | 6 months
  Effect of detection rate of early cancer and precancerous lesions on upper gastrointestinal tract from senior, intermediate and primary endoscopist with assistance of AQCS.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (6):
- China (6):
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Linyi People's Hospital, Dezhou, Shandong
  - Central Hospital of Shengli Oilfield, Dongying, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - PKUcare Luzhong Hospital, Zibo, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong

REFERENCES:
- [Derived] Zhou R, Liu J, Zhang C, Zhao Y, Su J, Niu Q, Liu C, Guo Z, Cui Z, Zhong X, Zhao W, Li J, Zhang X, Wang H, Sun S, Ma R, Chen X, Xu X, Zhu Y, Li Z, Zuo X, Li Y. Efficacy of a real-time intelligent quality-control system for the detection of early upper gastrointestinal neoplasms: a multicentre, single-blinded, randomised controlled trial. EClinicalMedicine. 2024 Aug 30;75:102803. doi: 10.1016/j.eclinm.2024.102803. eCollection 2024 Sep. PMID 39281103